CLINICAL TRIAL: NCT00136851
Title: A 6-Week Multi-center, Randomized, Double-Blind, Parallel Group Study Comparing the Efficacy of Amlodipine Besylate/Benazepril Versus Amlodipine in the Treatment of Severe Hypertension
Brief Title: Study Comparing the Efficacy of Amlodipine Besylate/Benazepril Versus Amlodipine in the Treatment of Severe Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCIB002FUS19
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2006-06

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — benazepril

INTERVENTIONS:
Drug: amlodipine besylate/benazepril hydrochloride

SUMMARY:
This trial is designed to study the efficacy of an amlodipine besylate/benazepril treatment regimen versus an amlodipine treatment regimen in the treatment of severe hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe hypertension

Exclusion Criteria:

* Diastolic blood pressure (DBP) < 60 mm Hg
* Serum potassium < 3.5 or > 5.5 mEq/L in the absence of all potassium supplements
* Refractory hypertension defined as systolic blood pressure (SBP) ≥ 180 mmHg and/or DBP ≥ 110 mmHg and unresponsive to triple-drug regimens

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2004-12; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving blood pressure goal which is defined as < 140/90 mm Hg, or < 130/80 mm Hg in subjects with diabetes after 4 weeks

SECONDARY OUTCOMES:
Percentage of subjects achieving blood pressure goal, defined as < 140/90 mm Hg, or < 130/80 mm Hg in subjects with diabetes after 6 weeks
Change from baseline in the mean sitting systolic blood pressure after 4 and 6 weeks
Change from baseline in the mean sitting diastolic blood pressure after 4 and 6 weeks
Percentage of subjects with swelling in legs or arms after 4 and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Izzo JL Jr, Purkayastha D, Hall D, Hilkert RJ. Comparative efficacy and safety of amlodipine/benazepril combination therapy and amlodipine monotherapy in severe hypertension. J Hum Hypertens. 2010 Jun;24(6):403-9. doi: 10.1038/jhh.2009.80. Epub 2009 Nov 5. PMID 19890370